CLINICAL TRIAL: NCT06728267
Title: Effects of Core Stabilization Training on Trunk Muscle Endurance, Respiratory Function and Quality of Life in Child and Adolescent Underwater Rugby Athletes
Brief Title: Core Stabilization Training in Child and Adolescent Underwater Rugby Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ozden Gokcek (Other)
Responsible Party: Sponsor-Investigator, Ozden Gokcek, Principal Investigator, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/12
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Core Stabilization; Trunk Muscle Endurance; Respiratory Function; Quality of Life
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will receive core stabilization training in addition to the training process. This training will be given for 6 weeks, 3 days a week, with 2 sets of 10 repetitions for the first two weeks, 2 sets of 15 repetitions for the second two weeks, and 3 sets of 12 repetitions for the third two weeks.
  Interventions: Other: Core stabilization training; Other: Training
- Control Group (Active Comparator): The control group will be monitored throughout the training period and will not be given any training program.
  Interventions: Other: Training

INTERVENTIONS:
Other: Core stabilization training — Exercise training will be given for 6 weeks, 3 days a week, 2 sets of 10 repetitions for the first two weeks, 2 sets of 15 repetitions for the second two weeks, and 3 sets of 12 repetitions for the third two weeks.
  Arms: Experimental Group
Other: Training — Routine training sessions conducted by coaches specific to the sport of underwater rugby.

SUMMARY:
Demographic information of children aged 9-17 who volunteer to participate in the study and who play underwater rugby will be recorded, and all participants; respiratory function will be assessed with a portable spirometer (Cosmed Poni FX) device, respiratory muscle strength will be assessed with a portable (micro RPM brand) electronic mouth pressure measurement device, and quality of life will be assessed with the KIDSCREEN scale. Core muscle endurance will be assessed with trunk flexion, trunk extension, lateral plank tests and flat plank test developed by McGill.

Respiratory muscle strength will be measured according to ATS/ERS criteria using a portable electronic mouth pressure measurement device (micro RPM brand). Respiratory function test will be performed using a portable spirometer (Cosmed Pony FX) to assess respiratory function. Capillary blood oxygen saturation of children will be recorded according to pulse oximetry results. Blood pressure will be measured with a cuff of appropriate size after a 5-minute rest according to age, gender and height percentile.

The experimental group will receive core stabilization training in addition to the training process. This training; Exercise training will be provided for 6 weeks, 3 days a week, 2 sets of 10 repetitions for the first two weeks, 2 sets of 15 repetitions for the second two weeks, and 3 sets of 12 repetitions for the third two weeks (Rahmat, et al., 2014). MIP/MEP values will be evaluated once a week. The control group will be monitored during the training and no training program will be given. The exercise program will be applied at the end of the project by being included in the follow-up list. The children will be taken to the second evaluation 6 weeks after the first evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Doing underwater rugby.
* No mental problems.
* Able to cooperate.

Exclusion Criteria:

* Diagnosed with respiratory system disease.
* Kyphoscoliosis and/or advanced postural alignment problems that will affect respiratory function.
* Any orthopedic and neurological problems.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Trunk Extension Test | At the beginning and at the end of 6 weeks of exercise.
  The time it takes to remain in a face down position on a stretcher, with ankles and knees fixed on the stretcher, the body outside the edge of the stretcher and 25 cm above the ground, with hands crossed in front, holding the shoulders without changing position, will be recorded in seconds.
Trunk Flexion Test | At the beginning and at the end of 6 weeks of exercise.
  The time spent in sit-up position on the floor mat, with the trunk upright at a 60-degree angle, knees and hips in a 90-degree flexion position, feet supported by the assistant and fixed on the ground, hands crossed on the chest, without changing position will be recorded in seconds.
Lateral Plank Test | At the beginning and at the end of 6 weeks of exercise.
  The time spent in the lateral plank position, with one foot supported on the other, straight along the body length, hips up, one elbow supporting the ground, the other holding the crossed shoulder in front, without changing position will be recorded in seconds.
Straight Plank Test | At the beginning and at the end of 6 weeks of exercise.
  The time it takes to remain in the push-up position, with the fingertips on the ground, the elbows bent and touching the ground, and the hips up without changing position will be recorded in seconds.
Muscle Strength | At the beginning and at the end of 6 weeks of exercise.
  According to the muscle test method found by Dr. Lovett, the muscle strength test is performed by scoring 0-5. Abdominal muscles, oblique trunk flexors and back extensors will be tested for muscle strength. Two separate tests will be performed for the lower and upper parts of the abdominal muscles.
Evaluation of the Stabilizing Function of the Transversus Abdominis Muscle | At the beginning and at the end of 6 weeks of exercise.
  Abdominal muscle activity was measured using the pressure biofeedback unit (PBU) during abdominal inhalation maneuver in the prone position and during posterior pelvic tilt movement in the supine position. Transversus abdominis muscle activity is assessed using the PBU with abdominal inhalation maneuver in the prone position. The cuff of the BBU is placed between the midpoint of the line connecting both spina iliaca anterior superiors of the participant and the umbilical cord. The participant is asked to breathe comfortably abdominally. The valve of the manometer is closed and the cuff is inflated to a pressure of 70 mmHg. All participants are given the standard command of "pull your abdomen in without moving your spine and hips and wait 10 seconds". The amount of pressure decrease in the manometer is recorded. The measurement will be repeated 3 times with 2-minute rest periods to prevent possible muscle fatigue and the average will be taken.
Respiratory Muscle Strength | At the beginning and at the end of 6 weeks of exercise.
  Respiratory muscle strength will be measured using a portable electronic mouth pressure measuring device (micro RPM brand) according to ATS/ERS criteria. Maximal inspiratory pressure (MIP) will be measured at residual volume and during deep inspiration. Maximal expiratory pressure (MEP) will be measured at total lung capacity and during deep expiration. Tests will be performed in the sitting position using a nose clip. Inspiratory and expiratory muscle strength values will be expressed as a percentage of the expected value.
Respiratory Function Test | At the beginning and at the end of 6 weeks of exercise.
  Respiratory function test will be performed using a portable spirometer (Cosmed Pony FX). The test will be performed in a sitting position, with the patient first asked to take a deep breath and then exhale quickly through the spirometer. A nose clip will be used during exhalation. Forced vital capacity (FVC), forced expiratory volume in one second (FEV1), FEV1/FVC will be recorded. Respiratory function test parameters will be expressed as a percentage of expected values according to age, height, body weight and sex.
Saturation | At the beginning and at the end of 6 weeks of exercise.
  Capillary blood oxygen saturation will be determined by pulse oximetry.
Blood Pressure | At the beginning and at the end of 6 weeks of exercise.
  ssessment of blood pressure is important to detect hypertension or hypovolemic shock. A blood pressure value in the 50th percentile for a child's age, gender, and height is considered the midpoint of the normal range. A reading above the 95th percentile indicates hypertension.
KIDSCREEN Health-Related Quality of Life Questionnaire | At the beginning and at the end of 6 weeks of exercise.
  KIDSCREEN52, which has been validated and reliable in Turkish, is a general purpose quality of life scale developed for children and adolescents aged 8-18, consisting of 52 questions in total. The KIDSCREEN-27 short form is a scale consisting of 27 questions and 5 dimensions, taken from KIDSCREEN-52. KIDSCREEN-27 consists of the dimensions of physical well-being (5 items), psychological well-being (7 items), autonomy and relationships with parents (7 items), social support and peers (4 items) and school environment (4 items).

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)